CLINICAL TRIAL: NCT03881332
Title: Clinical Observational Study Using Iohexol to Measure Perioperative Glomerular Filtration Rate in Patients Undergoing Robotic Surgery for Rectum or Large Bowel Cancers
Brief Title: Measurement of Perioperative Glomerular Filtration Rate
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Lars Marius Ytrebo, Professor, University Hospital of North Norway
Other Study IDs: 2018/1934
Record Dates: First submitted 2019-03-16; First posted 2019-03-19 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Rectal Cancer; Colon Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to monitor glomerular filtration rate (GFR)during the perioperative phase of patients undergoing robotic surgery for rectum or large bowel cancers. We will use both a single injection and a continuous infusion of iohexol to measure kidney function for 72 hours after surgery.

DETAILED DESCRIPTION:
The considerable morbidity and mortality associated with perioperative acute kidney injury (AKI) is well documented and known to complicate recovery from surgery.

Accurate, direct measurements of glomerular filtration rate (GFR) may provide a tool to monitor perioperative onset of rapidly changing renal function. This may subsequently lead to design of randomized controlled trials examining the effects of earlier intervention with the aim to reduce the incidence of perioperative AKI.

Recently a protocol for continuous infusion of low-dose iohexol (CILDI) as a measure of GFR in stable patients over a range of GFR (28-128 mL/min/1.73 m2) has been developed. Accuracy of this infusion protocol was confirmed with the single bolus injection (SBI) method. Data also showed that the continuous infusion protocol of low-dose iohexol is an accurate and precise method when measuring changing GFR even in critical ill patients with variable AKI risks. Accordingly, SBI and CILDI together now allow us to explore unanswered research questions related to perioperative change in renal function.

ELIGIBILITY:
Inclusion Criteria:

* Rectum or colon cancer

Exclusion Criteria:

* Acute kidney injury grade 3 or higher

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive elective rectum and colonic cancer patients due for robot surgery
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate | 72 hours
  Measured glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Lars Marius Ytrebo, PhD, Study Chair — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway